CLINICAL TRIAL: NCT00796835
Title: Dose-proportionality Study of the Five ER OROS Paliperidone To-be-marketed Tablet Strengths (3, 6, 9, 12, and 15 mg) in Healthy Male Subjects
Brief Title: A Dose-proportionality Study of Five Tablet Strengths of ER OROS Paliperidone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR004210
Record Dates: First submitted 2008-11-20; First posted 2008-11-24 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2010-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Mood disorders; Antipsychotic drugs; ER OROS Paliperidone
MeSH Terms: conditions — Schizophrenia; Mood Disorders

INTERVENTIONS:
Drug: ER OROS Paliperidone

SUMMARY:
The purpose of this study is to evaluate the dose proportionality of the 3-, 6-, 9-, 12-, and 15-mg tablets of ER OROS paliperidone. Additionally, the safety and tolerability of the treatments in healthy volunteers will be assessed.

DETAILED DESCRIPTION:
This study is designed as a single-center, open-label, randomized, 5 treatment-period, crossover study in healthy male adults. The study consists of a screening phase and an open-label treatment phase during which each volunteer will receive 5 treatments of study drug in a random order and separated by a washout period of 10 to 14 days. Treatments will consist of a single oral dose of: A) 1 tablet containing 3 mg ER OROS paliperidone; B) 1 tablet containing 6 mg ER OROS paliperidone; C) 1 tablet containing 9 mg ER OROS paliperidone; D) 1 tablet containing 12 mg ER OROS paliperidone; E) 1 tablet containing 15 mg ER OROS paliperidone. All treatments will be administered after an overnight fast. Volunteers are to remain in bed for 4 hours after dosing and are strongly advised to remain in bed for up to 36 hours. Five different ER OROS paliperidone tablet strengths (3, 6, 9, 12, and 15 mg) will be developed with the intent to market. Since ER OROS paliperidone is an extended release formulation, this study is designed to show dose-proportional pharmacokinetics of all these dose strengths. Safety and tolerability will be monitored throughout the study. Treatments will consist of a single oral dose of: A) 1 tablet containing 3 mg ER OROS paliperidone; B) 1 tablet containing 6 mg ER OROS paliperidone; C) 1 tablet containing 9 mg ER OROS paliperidone; D) 1 tablet containing 12 mg ER OROS paliperidone; E) 1 tablet containing 15 mg ER OROS paliperidone

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (weight [kg]/height [m²]) of 18 to 28 kg/m², inclusive
* Normotensive with supine (5 minutes) blood pressure between the range of 100 to 140 mmHg systolic, inclusive, and 60 to 90 mmHg diastolic, inclusive
* Healthy on the basis of a prestudy physical examination, medical history, ECG, and the laboratory results of serum chemistry, hematology and urinalysis performed within 21 days before the first dose. If the results of the serum chemistry, hematology or urinalysis testing are not within the laboratory's reference ranges the volunteer can be included only if the investigator judges that the deviations are not clinically significant
* For renal function tests, the values must be within the normal laboratory reference range.

Exclusion Criteria:

* Recent history of alcohol or substance abuse, a positive test result for the urine drug screen at screening or upon admittance to the testing facility or a positive result for the alcohol breath test upon admittance to the testing facility
* Relevant history or presence of any cardiovascular (including myocardial infarct or cardiac arrhythmia), respiratory, neurologic (including seizures), psychiatric, renal, hepatic, gastrointestinal (including surgeries, severe gastrointestinal narrowing, and malabsorption problems), endocrine, hematologic or immunologic disease
* History of any cancer, with the exception of basal cell carcinoma
* At screening, has a sustained decrease of >20 mmHg in systolic blood pressure or a decrease of >10 mmHg in diastolic blood pressure after standing for at least 2 minutes that is not associated with an increase of >15 beats per minute (bpm) in heart rate
* Bradycardia (heart rate <50 bpm) as determined by screening ECG
* History of a positive result for any of the serology tests (hepatitis B, C, and HIV)
* History of smoking or use of nicotine-containing substances within the last 2 months, as determined by medical history and/or volunteer's verbal report. Volunteers must agree to refrain from use throughout the study

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2004-07; Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the dose proportionality of the 3-, 6-, 9-, 12-, and 15-mg tablets of ER OROS paliperidone

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of the treatments in healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A dose-proportionality study of five tablet strengths of ER OROS paliperidone — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1083&filename=CR004210_CSR.pdf